CLINICAL TRIAL: NCT05151627
Title: Effectiveness of Kinesio Taping and Conventional Physical Therapy in the Management of Knee Osteoarthritis
Brief Title: The Effectiveness of Kinesio Taping in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tabuk (Other)
Responsible Party: Principal Investigator, Shahul Hameed Pakkir Mohamed, ASSISTANT PROFESSOR, University of Tabuk
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S-1440-0070
Record Dates: First submitted 2021-11-20; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee; Osteoarthritis; Kinesio taping; TENS; Stretching; Strengthening exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KINESIO TAPING AND CONVENTIONAL PHYSICAL THERAPY (Experimental): Application of Kinesio taping following Transcutaneous Electrical Nerve Stimulation and Knee Exercises
  Interventions: Procedure: KINESIO TAPING; Device: CONVENTIONAL PHYSICAL THERAPY
- CONVENTIONAL PHYSICAL THERAPY (Experimental): Application of Transcutaneous Electrical Nerve Stimulation and Knee Exercises
  Interventions: Device: CONVENTIONAL PHYSICAL THERAPY

INTERVENTIONS:
Procedure: KINESIO TAPING — Kinesio taping The patient is in a supine position with full knee flexion. Prior to application, the skin surface was cleaned. This technique involved the use of two Y-cut strips and two I-cut strips.
  Arms: KINESIO TAPING AND CONVENTIONAL PHYSICAL THERAPY
Device: CONVENTIONAL PHYSICAL THERAPY — Transcutaneous Electrical Nerve Stimulation TENS device settings, such as the frequency of 32-50 Hz, pulse width of 80 ms, and symmetrical biphasic waveform. The surface electrodes were placed on the medial and lateral superior borders of the patella, as well as the medial and lateral inferior borders of the patella.
  Exercise therapy program The total duration of each exercise session was about 50 minutes, including warm-up-10 minutes, resistance exercise-20 minutes, balance and stability exercise-10 minutes, lower-limb stretching exercise-5 minutes, and cool-down exercise-5 minutes. The same assigned physical therapist supervised all of the sessions.

SUMMARY:
Knee osteoarthritis is the most common kind of arthritis that occurs due to degeneration of the joint articular cartilage, producing pain, stiffness, and impaired movement. Kinesio taping is a simple and inexpensive therapeutic procedure that can help with knee osteoarthritis symptoms. Kinesio taping is a high-stretch elastic adhesive material that allows the treated area to have free mobility. This technique was preferred by physical therapists for knee osteoarthritis rehabilitation because of its positive effects, such as decreased pain and increased mobility and muscular performance.

ELIGIBILITY:
Inclusion Criteria:

* Complaining of knee pain but no serious knee injuries
* No Physical therapy treatment taken for the past 3 months
* Painful range of motion (ROM)
* Significant decrease in active and passive ROM.

Exclusion Criteria:

* Knee surgery within the last three months
* Neural, articular, or muscular conditions affecting lower limb function
* Systemic arthritic diseases

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
NUMERICAL PAIN RATING SCALE | 6 weeks
  The average pain intensity was measured during the past week, with zero representing no pain and ten representing the worst pain.
GONIOMETRIC MEASUREMENT OF KNEE RANGE OF MOTION | 6 weeks
  Both the knee flexion and extension ROM were measured while the subject was in a prone position. The measurement was done three times and the average result was obtained.
WESTERN ONTARIO AND MCMASTER UNIVERSITIES OSTEOARTHRITIS INDEX (WOMAC) | 6 weeks
  The questionnaire was developed to measure treatment outcomes in patients with lower extremity osteoarthritis, such as pain, stiffness, and difficulty, and it employs a scale to categorize the difficulties in activities of daily living. For individuals with hip and knee osteoarthritis, the WOMAC scale is a valid and reliable outcome measurement.
TIMED UP AND GO (TUG) TEST | 6 weeks
  The test combines static and dynamic balance to assess a person's mobility. Getting out of a chair, walking three meters, turning around, and returning to the chair to sit. The international research OA society recommends a series of physical function measures (five performance-based) for individual with hip or knee OA, including the TUG test.24 The aforementioned outcome parameters are measured at three-time intervals: 0-week, 3-week, and 6-week.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tabuk, Tabuk, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 3 MONTHS
Access Criteria: ON REQUEST